CLINICAL TRIAL: NCT03930615
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of Letermovir (LET) Prophylaxis When Extended From 100 Days to 200 Days Post-transplant in Cytomegalovirus (CMV) Seropositive Recipients (R+) of an Allogenic Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Extension of Letermovir (LET) From Day 100 to Day 200 Post-transplant for the Prevention of Cytomegalovirus (CMV) Infection in Hematopoietic Stem Cell Transplant (HSCT) Participants (MK-8228-040)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 8228-040; MK-8228-040 (Other: Merck Sharp & Dohme Corp.); 194797 (Registry Identifier: JAPIC-CTI); 2018-001038-17 (EudraCT Number)
Record Dates: First submitted 2019-04-26; First posted 2019-04-29 (Actual); Results first posted 2022-11-01 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Cytomegalovirus Infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Letermovir (Experimental): Participants who received HSCT transplant and 100 days of LET prophylaxis were randomized to an additional 100 days of LET (480 mg once daily alone or 240 mg once daily for participants on cyclosporin A) treatment.
  Interventions: Drug: Letermovir
- Placebo (Placebo Comparator): Participants who received HSCT transplant and 100 days of LET prophylaxis were randomized to an additional 100 days of placebo treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Letermovir — LET tablet or intravenous infusion at a total daily dose of 240 mg (when given with cyclosporin A) or 480 mg (when given alone).
  Other Names: PREVYMIS™, MK-8228
  Arms: Letermovir
Drug: Placebo — Placebo was administered as tablets matched to LET or as inactive (saline or dextrose) intravenous infusion.
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of letermovir (LET) versus placebo when cytomegalovirus (CMV) prophylaxis was extended from 100 days to 200 days post-transplant in CMV seropositive participants who received an allogenic hematopoietic stem cell transplant (HSCT). It was hypothesized that LET is superior to placebo in the prevention of clinically-significant CMV infection when LET prophylaxis is extended from 100 to 200 days.

ELIGIBILITY:
Inclusion Criteria:

* have documented positive CMV serostatus (CMV immunoglobulin G [IgG] seropositive) for recipient (R+) at the time of transplant
* has a history of allogeneic HSCT (bone marrow, peripheral blood stem cell, or cord blood transplant) within ~100 days prior to randomization
* has undetectable CMV deoxyribonucleic acid (DNA) or detectable/not quantifiable CMV DNA from a plasma sample collected within 14 days prior to randomization
* has received LET as primary prophylaxis that started within 28 days of HSCT and continued through Week 14 post-transplant (± 1 week) prior to randomization
* is at high risk of CMV disease, defined as meeting one or more of the following criteria:
* has a related donor with at least 1 mismatch at 1 of the specified 3 human leukocyte antigen (HLA) gene loci (HLA-A, B, or DR)
* has an unrelated donor with at least one mismatch at one of the specified four HLA gene loci (HLA-A, B, C, and DRB1)
* has a haploidentical donor
* has umbilical cord blood as the stem-cell source
* has ex-vivo T-cell-depleted grafts
* has received anti-thymocyte globulin
* has received alemtuzumab
* has graft versus host disease (GVHD) or other conditions, requiring the use of systemic prednisone (or equivalent) at a dose of ≥1 mg/kg of body weight per day within 6 weeks of randomization
* for female participants, is not pregnant or breastfeeding, and is either not a woman of childbearing potential (WOCBP) or is a WOBCP who agrees to use acceptable contraception during the treatment period and for ≥28 days after the last dose of study drug.

Exclusion Criteria:

* has a history of CMV end-organ disease or preemptive treatment therapy for CMV after HSCT prior to randomization
* has a history of >14 days total of LET interruption during the first 100 days post-transplant prior to randomization
* has suspected or known hypersensitivity to active or inactive ingredients of LET formulations
* has severe hepatic insufficiency defined as Child-Pugh Class C within 14 days prior to randomization.
* has serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5× the upper limit of normal (ULN) within 14 days prior to randomization
* has end-stage renal impairment with a creatinine clearance less than 10 mL/min, as calculated by the Cockcroft-Gault equation using serum creatinine within 14 days prior to randomization
* has both moderate hepatic insufficiency AND moderate-to-severe renal insufficiency
* has an uncontrolled infection on the day of enrollment
* requires mechanical ventilation or is hemodynamically unstable at the time of enrollment
* has a documented positive result for a human immunodeficiency virus antibody (HIV-Ab) test at any time prior to screening, or for hepatitis C virus antibody (HCV-Ab) with detectable HCV ribonucleic acid (RNA), or hepatitis B surface antigen (HBsAg) within 6 months prior to screening.
* has active solid tumor malignancies with the exception of localized basal cell or squamous cell skin cancer or the condition under treatment (eg, lymphomas)
* has received cidofovir or CMV immunoglobulin with 30 days prior to screening
* is currently participating or has participated in a study with an unapproved investigational compound, monoclonal antibody, or device within 28 days or 5× half-life of the investigational compound or monoclonal antibody, whichever is longer, of initial dosing in this study
* has previously participated in this study or any other study involving LET, or is currently participating in any study involving administration of a CMV vaccine or another CMV investigational agent, or is planning to participate in a study of a CMV vaccine or another CMV investigational agent during the course of this study
* is pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through 28 days after the last dose of study therapy
* is expecting to donate eggs starting from the time of consent through 28 days after the last dose of study therapy
* has clinically relevant drug or alcohol abuse within 12 months of screening that may interfere with participant treatment, assessment, or compliance with the protocol as assessed by the investigator
* has a history or current evidence of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or would be put at undue risk as judged by the investigator, such that it is not in the best interest of the participant to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (32):
- United States (10):
  - City of Hope National Medical Center ( Site 0158), Duarte, California
  - University of California Davis Medical Center ( Site 0156), Sacramento, California
  - University of Miami, Sylvester Comprehensive Cancer Center ( Site 0160), Miami, Florida
  - Indiana Blood and Marrow Transplantation ( Site 0175), Indianapolis, Indiana
  - Brigham & Women's Hospital ( Site 0161), Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Med Ctr ( Site 0174), Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center ( Site 0164), New York, New York
  - Duke University Medical Center ( Site 0169), Durham, North Carolina
  - The University of Texas MD Anderson Cancer Center ( Site 0154), Houston, Texas
  - Fred Hutchinson Cancer Research Center ( Site 0152), Seattle, Washington
- France (6):
  - Centre Hospitalier Universitaire Dupuytren ( Site 0182), Limoges, Haute-Vienne
  - Hopital Saint Eloi ( Site 0031), Montpellier, Herault
  - Centre Hopitalier Lyon Sud ( Site 0039), Pierre-Bénite, Rhone
  - CHU Henri Mondor ( Site 0032), Créteil, Val-de-Marne
  - Institut Gustave Roussy ( Site 0038), Villejuif, Val-de-Marne
  - CHU Hopital Saint Antoine ( Site 0036), Paris
- Germany (3):
  - Universitaetsklinikum Heidelberg-Medizinische Klinik V ( Site 0042), Heidelberg, Baden-Wurttemberg
  - Universitaetsklinik Koeln ( Site 0041), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Muenster ( Site 0043), Münster, North Rhine-Westphalia
- Italy (5):
  - ASST Spedali Civili di Brescia ( Site 0052), Brescia, Lombardy
  - IRCCS Ospedale San Raffaele ( Site 0051), Milan
  - Fondazione PTV Policlinico Tor Vergata ( Site 0054), Roma
  - Policlinico Umberto I ( Site 0056), Roma
  - Policlinico Universitario Agostino Gemelli ( Site 0055), Roma
- Japan (3):
  - Jichi Medical University Hospital ( Site 0123), Shimotsuke, Tochigi
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital ( Site 0121), Hiroshima
  - National Hospital Organization Kumamoto Medical Center ( Site 0122), Kumamoto
- United Kingdom (5):
  - Queen Elizabeth University Hospital [Glasgow, UK] ( Site 0096), Glasgow, Glasgow City
  - 1Kings College Hospital ( Site 0091), London, London, City of
  - UCL Cancer Institute ( Site 0093), London, London, City of
  - Manchester Royal Infirmary ( Site 0097), Manchester
  - Freeman Hospital Newcastle upon Tyne Foundation NHS Trust ( Site 0092), Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Russo D, Schmitt M, Pilorge S, Stelljes M, Kawakita T, Teal VL, Haber B, Bopp C, Dadwal SS, Badshah C. Efficacy and safety of extended duration letermovir prophylaxis in recipients of haematopoietic stem-cell transplantation at risk of cytomegalovirus infection: a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Haematol. 2024 Feb;11(2):e127-e135. doi: 10.1016/S2352-3026(23)00344-7. Epub 2023 Dec 21. PMID 38142695
- [Derived] Dwabe S, Hsiao M, Ali A, Rodman J, Savitala-Damerla L, Nazaretyan S, Kimberly Schiff NP, Tam E, Ladha A, Woan K, Chaudhary P, Yaghmour G. Real world experience: Examining outcomes using letermovir for CMV prophylaxis in high-risk allogeneic hematopoietic stem cell patients in the setting of using T-cell depletion as GVHD prophylaxis. Transpl Immunol. 2023 Feb;76:101769. doi: 10.1016/j.trim.2022.101769. Epub 2022 Dec 2. PMID 36464218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cytomegalovirus (CMV)-seropositive recipients (R+) of a hematopoietic stem cell transplant (HSCT) who had received letermovir (LET) prophylaxis through Week 14 (~100 days) post-transplant and were at high risk for CMV infection and/or disease were enrolled in this study.
Period: Overall Study
Arm/Group | Letermovir | Placebo
Started (Randomized) | 145 | 75
Treated | 144 | 74
Completed | 118 | 63
Not Completed | 27 | 12
Not completed — Death | 9 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 3 | 4
Not completed — Withdrawal by Subject | 13 | 2
Not completed — Not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Letermovir | Placebo | Total
Number analyzed (Participants) | 144 | 74 | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (14.3) | 52.7 (12.9) | 52.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 31 | 83
  Male | 92 | 43 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 106 | 53 | 159
  Unknown or Not Reported | 25 | 13 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 8 | 24
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 3 | 1 | 4
  White | 113 | 60 | 173
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 8 | 4 | 12
Donor Stratum [Count of Participants; unit: Participants]
  Haploidentical | 45 | 22 | 67
  Non-haploidentical | 99 | 52 | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Significant CMV Infection From Week 14 (~100 Days) Post-transplant Through Week 28 (~200 Days) Post-transplant
Description: Clinically significant CMV infection is either the onset of probable or proven CMV end-organ disease or initiation of anti-CMV preemptive therapy (PET) with approved anti-CMV agents (ganciclovir, valganciclovir, foscarnet, and/or cidofovir) based on documented CMV viremia and the clinical condition of the participant. Missing values were handled by the observed failure (OF) approach where failure was defined as all participants who develop clinically significant CMV infection or discontinue prematurely from the study with CMV viremia from week 14 (~100 days) through week 28 post-transplant. It was hypothesized that LET is superior to placebo in the prevention of clinically significant CMV infection when LET prophylaxis is extended from 100 to 200 days.
Time Frame: From Week 14 post-transplant to Week 28 post-transplant (approximately 14 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 2.8 | 18.9
Statistical Analysis 1: Comparison: Letermovir vs Placebo; It was hypothesized that LET is superior to placebo in the prevention of clinically significant CMV infection; Test type: Superiority; p = 0.0005, Mantel Haenszel — A one-sided p-value ≤0.0249 was used for declaring statistical significance; Stratum adjusted; Treatment Difference = -16.1, 95% CI 2-sided [-25.8 to -6.5] — Letermovir minus placebo; 95% CIs for the treatment differences in percent response were calculated using stratum adjusted Mantel Haenszel method with the difference weighted by the harmonic mean of sample size per arm for each stratum (haploidentical donor yes or no)

2. Secondary Outcome: Percentage of Participants Experiencing ≥1 Adverse Events (AEs) From Week 14 (~100 Days) Post-transplant Through Week 28 (~200 Days) Post-transplant
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: From Week 14 post-transplant to Week 28 post-transplant (approximately 14 weeks)
Population: All randomized participants who received at least 1 dose of study intervention according to the study intervention they received.
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 88.9 | 93.2
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Other; Difference in Percentage = -4.4, 95% CI 2-sided [-11.8 to 4.7] — Letermovir minus Placebo; Miettinen & Nurminen method

3. Secondary Outcome: Percentage of Participants Withdrawing From Study Drug Due to an AE From Week 14 (~100 Days) Post-transplant Through Week 28 (~200 Days) Post-transplant
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: From Week 14 post-transplant to Week 28 post-transplant (approximately 14 weeks)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 4.9 | 1.4
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Other; Difference in Percentage = 3.5, 95% CI 2-sided [-2.7 to 8.6] — Letermovir minus Placebo; Miettinen & Nurminen method

4. Secondary Outcome: Percentage of Participants With Clinically Significant CMV Infection From Week 14 Post-transplant Through Week 38 Post-transplant
Description: Clinically significant CMV infection is either the onset of probable or proven CMV end-organ disease or initiation of anti-CMV PET with approved anti-CMV agents (ganciclovir, valganciclovir, foscarnet, and/or cidofovir) based on documented CMV viremia and the clinical condition of the participant. Missing values were handled by the OF approach where failure was defined as all participants who develop clinically significant CMV infection or discontinue prematurely from the study with CMV viremia from week 14 (~100 days) through week 38 post-transplant.
Time Frame: From Week 14 post-transplant to Week 38 post-transplant (approximately 24 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 14.6 | 20.3
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority; p = 0.1591, Mantel Haenszel; Stratum adjusted; Treatment Difference = -5.7, 95% CI 2-sided [-16.8 to 5.4] — Letermovir minus placebo; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With Clinically Significant CMV Infection From Week 14 Post-transplant Through Week 48 Post-transplant
Description: Clinically significant CMV infection is either the onset of probable or proven CMV end-organ disease or initiation of anti-CMV PET with approved anti-CMV agents (ganciclovir, valganciclovir, foscarnet, and/or cidofovir) based on documented CMV viremia and the clinical condition of the participant. Missing values were handled by the OF approach where failure was defined as all participants who develop clinically significant CMV infection or discontinue prematurely from the study with CMV viremia from week 14 (~100 days) through week 48 post-transplant.
Time Frame: From Week 14 post-transplant to Week 48 post-transplant (approximately 34 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 14.6 | 20.3
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority; p = 0.1591, Mantel Haenszel; Stratum adjusted; Treatment Difference = -5.7, 95% CI 2-sided [-16.8 to 5.4] — Letermovir minus placebo; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Time to Onset of Clinically Significant CMV Infection From Week 14 Post-transplant to Week 28 Post-transplant
Description: Clinically significant CMV infection is either the onset of probable or proven CMV end-organ disease or initiation of anti-CMV PET with approved anti-CMV agents (ganciclovir, valganciclovir, foscarnet, and/or cidofovir) based on documented CMV viremia and the clinical condition of the participant. Time to onset of clinically significant CMV infection is the elapsed time from transplant to the onset of CMV end-organ disease or to the initiation of anti-CMV PET. Time to onset was determined from the Kaplan-Meier method for censored data.
Time Frame: From Week 14 post-transplant to Week 28 post-transplant (approximately 14 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Days | NA [NA to NA] — NA means that due to the less than 50% incidence of clinically significant CMV infection, the median time was not reached. | NA [NA to NA] — NA means that due to the less than 50% incidence of clinically significant CMV infection, the median time was not reached.

7. Secondary Outcome: Time to Onset of Clinically Significant CMV Infection From Week 14 Post-transplant to Week 48 Post-transplant
Description: as for outcome 6
Time Frame: From Week 14 post-transplant to Week 48 post-transplant (approximately 34 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Days | NA [NA to NA] — NA means that due to the less than 50% incidence of clinically significant CMV infection, the median time was not reached. | NA [NA to NA] — NA means that due to the less than 50% incidence of clinically significant CMV infection, the median time was not reached.

8. Secondary Outcome: Percentage of Participants With CMV Viremia Who Started PET From Week 14 Post-transplant to Week 28 Post-transplant
Description: The percentage of participants with CMV viremia who initiated PET of anti-CMV agents (ganciclovir, valganciclovir, foscarnet, and/or cidofovir) was determined. Missing values were handled with the OF approach, where failure was defined as all participants who develop clinically significant CMV infection or discontinue prematurely from the study with CMV viremia from week 14 through week 28 post-transplant.
Time Frame: From Week 14 post-transplant to Week 28 post-transplant (approximately 14 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 2.1 | 16.2
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority; p = 0.0012, Mantel Haenszel; Stratum adjusted; Treatment difference = -14.1, 95% CI 2-sided [-23.3 to -5.0] — Letermovir minus placebo; [other analysis details as in outcome 1, analysis 1]

9. Secondary Outcome: Percentage of Participants With CMV Viremia Who Started PET From Week 14 Post-transplant to Week 48 Post-transplant
Description: The percentage of participants with CMV viremia who initiated PET of anti-CMV agents (ganciclovir, valganciclovir, foscarnet, and/or cidofovir) was determined. Missing values were handled with the OF approach, where failure was defined as all participants who develop clinically significant CMV infection or discontinue prematurely from the study with CMV viremia from week 14 through week 48 post-transplant.
Time Frame: From Week 14 post-transplant to Week 48 post-transplant (approximately 34 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 13.2 | 18.9
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority; p = 0.1494, Mantel Haenszel; Stratum adjusted; Treatment Difference = -5.7, 95% CI 2-sided [-16.5 to 5.1] — Letermovir minus placebo; [other analysis details as in outcome 1, analysis 1]

10. Secondary Outcome: Percentage of Participants With All-cause Mortality From Week 14 Post-transplant to Week 28 Post-transplant
Description: The percentage of participants who died due to any cause (all-cause mortality) from Week 14 to Week 28 was determined.
Time Frame: From Week 14 post-transplant to Week 28 post-transplant (approximately 14 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 2.1 | 1.4
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority; p = 0.6244, Mantel Haenszel; Stratum adjusted; Treatment difference = 0.7, 95% CI 2-sided [-3.8 to 5.3] — Letermovir minus placebo; [other analysis details as in outcome 1, analysis 1]

11. Secondary Outcome: Percentage of Participants With All-cause Mortality From Week 14 Post-transplant to Week 48 Post-transplant
Description: The percentage of participants who died due to any cause (all-cause mortality) from Week 14 to Week 48 was determined.
Time Frame: From Week 14 post-transplant to Week 48 post-transplant (approximately 34 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 8.3 | 8.1
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority; p = 0.5264, Mantel Haenszel; Stratum adjusted; Treatment Difference = 0.3, 95% CI 2-sided [-7.9 to 8.4] — Letermovir minus placebo; [other analysis details as in outcome 1, analysis 1]

12. Secondary Outcome: Time to All-cause Mortality From Week 14 Post-transplant to Week 28 Post-transplant
Description: Time to all-cause mortality is the time elapsed after Week 14 post-transplant and death due to any cause, and was determined from the Kaplan-Meier method for censored data.
Time Frame: From Week 14 post-transplant to Week 28 post-transplant (approximately 14 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Days | NA [NA to NA] — NA means that as participants were followed for less than a year after transplant, this was insufficient time to reach a median survival time. | NA [NA to NA] — NA means that as participants were followed for less than a year after transplant, this was insufficient time to reach a median survival time.

13. Secondary Outcome: Time to All-cause Mortality From Week 14 Post-transplant to Week 48 Post-transplant
Description: as for outcome 12
Time Frame: From Week 14 post-transplant to Week 48 post-transplant (approximately 34 weeks)
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 144 | 74
Days | NA [NA to NA] — NA means that as participants were followed for less than a year after transplant, this was insufficient time to reach a median survival time. | NA [NA to NA] — NA means that as participants were followed for less than a year after transplant, this was insufficient time to reach a median survival time.

ADVERSE EVENTS:
Time Frame: All-cause mortality: From 14 weeks post-transplant up to 48 weeks post-transplant (approximately 34 weeks); adverse events (AEs) and serious AEs (SAEs): From 14 weeks post-transplant up to 30 weeks post-transplant (approximately 16 weeks).
Description: The population analyzed for all-cause mortality (death due to any cause) was all randomized participants. The population analyzed for AEs was all randomized participants who received at least 1 dose of study intervention according to the study intervention they received. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Arm/Group | Letermovir | Placebo
All-Cause Mortality (participants affected / at risk) | 16/145 | 8/75
Serious Adverse Events (participants affected / at risk) | 49/144 | 27/74
Other Adverse Events (participants affected / at risk) | 100/144 | 58/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=144) | Placebo (N=74)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pure white cell aplasia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Aplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 1 (2)
Graft versus host disease (Immune system disorders) | 9 (9) | 6 (6)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Adenoviral haemorrhagic cystitis (Infections and infestations) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (4)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cerebral toxoplasmosis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Human herpesvirus 6 infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Myelitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Escherichia test positive (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 3 (3)
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral T-cell lymphoma unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=144) | Placebo (N=74)
Anaemia (Blood and lymphatic system disorders) | 8 (9) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 16 (19) | 11 (12)
Nausea (Gastrointestinal disorders) | 17 (19) | 15 (17)
Vomiting (Gastrointestinal disorders) | 9 (10) | 3 (4)
Fatigue (General disorders) | 5 (6) | 5 (5)
Oedema (General disorders) | 0 (0) | 4 (4)
Oedema peripheral (General disorders) | 12 (12) | 9 (10)
Pyrexia (General disorders) | 12 (13) | 9 (13)
Graft versus host disease (Immune system disorders) | 45 (61) | 22 (34)
Cytomegalovirus infection (Infections and infestations) | 3 (4) | 4 (4)
Cytomegalovirus infection reactivation (Infections and infestations) | 6 (6) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 5 (5)
Alanine aminotransferase increased (Investigations) | 5 (5) | 4 (5)
Neutrophil count decreased (Investigations) | 4 (4) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7) | 11 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Dizziness (Nervous system disorders) | 3 (3) | 4 (5)
Headache (Nervous system disorders) | 10 (11) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 9 (11) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (2):
  • Study Protocol (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03930615/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT03930615/SAP_001.pdf